CLINICAL TRIAL: NCT02561416
Title: Cost-utility and Biological Underpinnings of Mindfulness-Based Stress Reduction (MBSR) in Fibromyalgia Syndrome: A Three-arm Randomized, Controlled Trial (EUDAIMON Project)
Brief Title: Cost-utility and Biological Underpinnings of MBSR in Fibromyalgia Syndrome
Acronym: EUDAIMON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Carlos III Health Institute (Other Government); Preventive Services and Health Promotion Research Network (Other); Parc Sanitari Sant Joan de Déu (Other)
Responsible Party: Principal Investigator, Juan Vicente Luciano, PhD, Fundació Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP14/00087; PI15/00383 (Other Grant/Funding Number: Institute of Health Carlos III)
Record Dates: First submitted 2015-09-23; First posted 2015-09-28 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia syndrome; Mindfulness (MBSR); Neuroimaging; Cytokines; Randomized Controlled Trial; Cost-effectiveness; Psychoeducation (FibroQol)
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mindfulness-Based Stress Reduction (Experimental): Mindfulness-Based Stress Reduction (MBSR) The MBSR consists in eight 2-h group sessions and an all-day mindfulness retreat, and offers intensive and structured training in mindfulness meditation to help patients to relate to their physical and psychological conditions in more accepting and nonjudgmental ways. Participants will be encouraged to engage in home mindfulness practices. Sessions will be lead by 4 MBSR accredited instructors.
  Interventions: Behavioral: MBSR; Drug: TAU
- Psycho-educational Program (Active Comparator): Psycho-educational Program (FibroQol) It consists of eight 2-h group sessions including information about FMS (4 sessions) based on a consensus document of the Health Department of Catalonia + autogenic relaxation (4 sessions).
  Interventions: Behavioral: FibroQol; Drug: TAU
- Treatment As Usual (Other): Treatment As Usual.
  Interventions: Drug: TAU

INTERVENTIONS:
Behavioral: MBSR — Session 1: Recognising the present moment Session 2: Engaging with the breath Session 3: Practice, practice, practice Session 4: Stress and the flow of emotions Session 5: Stress and thoughts: finding another place to stand Session 6: Interpersonal mindfulness / mindful communication. Session 7: Applying mindfulness Session 8: Making mindfulness a part of your life
  Arms: Mindfulness-Based Stress Reduction
Behavioral: FibroQol — Session 1: General information. Expectations of the patients. History of the illness. Principal and secondary symptoms in FM. Physiological mechanisms involved in the genesis of pain.
  Session 2: Relaxation training-I. Session 3: Diagnosis. Pharmacological and non-pharmacological treatments. Prognosis. Current model of health care in Catalonia. Units specialized in the treatment of FM.
  Session 4: Relaxation training-II. Session 5: Strategies to increase self-esteem and regulate emotions. Pain experience and recurrent invalidation. Social support (family and friends).
  Session 6: Relaxation training-III Session 7: Benefits of physical exercise in FM. Session 8: Relaxation training-IV.
  Arms: Psycho-educational Program
Drug: TAU — In Spain the treatment as usual provided in FMS is mainly pharmacological and adjusted to the symptomatic profile of the patient. Counselling about aerobic exercise adjusted to patients' physical limitations is usually also provided.
  Other Names: Usual care

SUMMARY:
Purpose:

Fibromyalgia syndrome (FMS) is a disabling condition mainly characterized by chronic widespread pain, disturbed sleep, fatigue, and distress. The estimated overall prevalence of FMS in Europe is 2.9% and it incurs in high personal, social and healthcare costs. Available treatments in FMS are not curative and there is some evidence of positive effects of mindfulness-based stress reduction (MBSR) in patients with chronic pain and FMS. Nevertheless, although promising, the positive findings obtained in previous studies implementing mindfulness-based interventions in patients with FMS have to be interpreted with caution due to important methodological limitations (e.g. absence of randomization, high attrition rates, or small sample sizes). Therefore, further research in larger studies using more adequate methodologies is warranted. Furthermore, little is known about putative neurobiological processes underpinning the effects of mindfulness training in patients with chronic pain.

Aims: The aim of this randomized, controlled trial (RCT) is two-fold: firstly, to assess the effectiveness and cost-utility of MBSR added to treatment as usual (TAU); and secondly, to evaluate the effects of the compared interventions on neurobiological parameters. Specifically, MBSR will be compared to an active control which was previously reported as a cost-effective intervention (TAU + FibroQol psycho-educational program; Luciano et al., 2013) and also vs. TAU alone (in a 12-month follow-up RCT). Brain structure and function of pain-relevant areas and levels of inflammation markers (cytokines) will be assessed pre-post interventions in half of the study participants.

Methods:

Design: RCT with three arms:

1. TAU + MBSR,
2. TAU + FibroQoL and
3. TAU.

Sample: 180 adults with FMS according to the ACR 1990 criteria (N=60 for each study arm) will be recruited from from the Parc Sanitari Sant Joan de Déu Rheumatology Service, Sant Boi de Llobregat, Spain. Half of the participants will be randomly selected to participate in the neurobiological pre-post evaluation (N= 30 each group). All patients will be assessed at baseline, post-intervention and 12-month follow-up for clinical variables, prep-post intervention for biomarkers study, and baseline and 12-month follow-up for cost-related variables.

DETAILED DESCRIPTION:
Detailed description of the study protocol has been published elsewhere (in an open-access journal):

http://bmccomplementalternmed.biomedcentral.com/articles/10.1186/s12906-016-1068-2

ELIGIBILITY:
General Inclusion Criteria:

* Patients of both genders between 18-65 years old.
* Verified diagnosis of FMS according to the American College of Rheumatology criteria (ACR 1990).
* Ability to understand Spanish language.
* Written informed consent.

General Exclusion Criteria:

* Participation in other clinical trials
* Cognitive impairment according to MINI (total score ≤ 24)
* Receiving psychological treatment during the last or the current year
* Previous experience with meditation or mind-body therapies.
* Physical/psychiatric comorbidity that interferes with treatment (any severe medical illness, psychotic symptoms, substance abuse).
* Not being able to attend to group sessions.
* Being involved in ongoing litigation relating to the FMS.

Additional Inclusion Criteria for the biomarkers sub-study (90 participants in total):

* Female gender
* Right-handed

Additional Exclusion Criteria for the biomarkers sub-study:

* Neoplastic illnesses (diagnosed from the medical history), infection, cardiopulmonary, vascular or other internal medical conditions
* Use of oral or local corticosteroids or anti-cytokine therapy
* Needle-phobia
* Impossibility of being scanned in MRI (due to agoraphobia, metal implants, pace-marker…)
* BMI> 36kg/m2 or >110Kg
* Consuming > 8 caffeine units per day
* Smoking > 5 cigarettes per day
* Acute pain not related to the FMS at the day of biomarkers evaluation
* Being pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness Evaluation: Revised Fibromyalgia Impact Questionnaire (FIQR) | Change from baseline scores at 12 months
Cost-utility: Client Service Receipt Inventory (CSRI) | Change from baseline scores at 12 months
Inflammatory markers: pro- and anti-inflammatory cytokines & hs-CRP | Change from baseline values at 2 months
EuroQoL questionnaire (EQ-5D-5L) | Change from baseline scores at 12 months
Structural neuroimaging: Voxel-Based Morphometry (VBM) | Change from baseline brain gray matter concentration at 2 months
  Analysis of morphometric changes associated with participation in the three study arms voxel-by-voxel across the brain and in functionally-defined brain regions of interest relating to meta-awareness, body awareness, memory consolidation-reconsolidation, and emotion regulation.
Functional neuroimaging: pulsed continuous arterial spin labeling (pCASL) | Change from baseline regional cerebral blood flow at 2 months
  Analysis of changes in regional cerebral blood flow representing response to treatment throughout the brain and in a priori-specified network of brain regions postulated to underpin the sensory-discriminative, cognitive-evaluative and affective-motivational aspects of the pain experience.

SECONDARY OUTCOMES:
Hamilton Anxiety and Depression Scale (HADS) | Baseline, 2-month & 12-month follow-up
Perceived Stress Scale (PSS-10) | Baseline, 2-month & 12-month follow-up
Multidimensional Inventory of Subjective Cognitive Impairment (MISCI) | Baseline, 2-month & 12-month follow-up
Pain Catastrophising Scale (PCS) | Baseline, 2-month & 12-month follow-up
Fibromyalgia Survey Diagnostic Criteria (FSDC) | Baseline, 2-month & 12-month follow-up

OTHER OUTCOMES:
Five Facets Mindfulness Questionnaire (FFMQ) | Baseline, 2-month & 12-month follow-up
  Process variable
Self-Compassion Scale (SCS-12) | Baseline, 2-month & 12-month follow-up
  Process variable
Psychological Inflexibility in Pain Scale (PIPS) | Baseline, 2-month & 12-month follow-up
  Process variable
Checklist - Adverse events of the interventions | 2-month
  Control variable
Credibility/Expectancy Questionnaire (CEQ) | Baseline (MBSR & FibroQol groups)
  Control variable
Mini-Mental State Examination (MMSE) | Baseline
  Screening measure
Structured Clinical Interview for DSM Axis I Disorders (SCID-I) | Baseline
  Screening measure

CONTACTS AND LOCATIONS:
Overall Officials: Juan V. Luciano, PhD, Principal Investigator — Teaching, Research & Innovation Unit - Parc Sanitari Sant Joan de Déu
Locations (1):
- Teaching, Research & Innovation Unit - Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medina S, O'Daly OG, Howard MA, Feliu-Soler A, Luciano JV. Differential Brain Perfusion Changes Following Two Mind-Body Interventions for Fibromyalgia Patients: an Arterial Spin Labelling fMRI Study. Mindfulness (N Y). 2022;13(2):449-461. doi: 10.1007/s12671-021-01806-2. Epub 2022 Jan 5. PMID 35222735
- [Derived] Perez-Aranda A, Feliu-Soler A, Montero-Marin J, Garcia-Campayo J, Andres-Rodriguez L, Borras X, Rozadilla-Sacanell A, Penarrubia-Maria MT, Angarita-Osorio N, McCracken LM, Luciano JV. A randomized controlled efficacy trial of mindfulness-based stress reduction compared with an active control group and usual care for fibromyalgia: the EUDAIMON study. Pain. 2019 Nov;160(11):2508-2523. doi: 10.1097/j.pain.0000000000001655. PMID 31356450
- [Derived] Feliu-Soler A, Borras X, Penarrubia-Maria MT, Rozadilla-Sacanell A, D'Amico F, Moss-Morris R, Howard MA, Fayed N, Soriano-Mas C, Puebla-Guedea M, Serrano-Blanco A, Perez-Aranda A, Tuccillo R, Luciano JV. Cost-utility and biological underpinnings of Mindfulness-Based Stress Reduction (MBSR) versus a psychoeducational programme (FibroQoL) for fibromyalgia: a 12-month randomised controlled trial (EUDAIMON study). BMC Complement Altern Med. 2016 Feb 27;16:81. doi: 10.1186/s12906-016-1068-2. PMID 26921267